CLINICAL TRIAL: NCT03603275
Title: Assessing Hemophilia A Patient and Physician Reasons and Expectations for Switching Treatment to Kovaltry & Jivi: A Nested Study Within an Existing Registry
Brief Title: Assessing Physician and Hemophilia A Patient Reasons and Expectations for Switching Treatment to Kovaltry & Jivi: A Nested Study Within an Existing Registry
Status: Terminated | Type: Observational
Why Stopped: Insufficient data
Sponsor: Bayer (Industry)
Collaborators: American Thrombosis and Hemostasis Network (Network)
Responsible Party: Sponsor
Other Study IDs: 19866
Record Dates: First submitted 2018-07-20; First posted 2018-07-27 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient/caregiver of Kovaltry or Jivi: Patients who are switching factor replacement products to Kovaltry or Jivi and patients who have switched factor replacement products to Kovaltry or Jivi previously
  Interventions: Drug: New FVIII products
- Physician Group: Physicians participating in the study are associated with US hemophilia treatment centers that are affiliated with the ATHN hemophilia treatment center network

INTERVENTIONS:
Drug: New FVIII products — Kovaltry or Jivi prescribed by the treating Physician
  Groups: Patient/caregiver of Kovaltry or Jivi

SUMMARY:
This US study aims to assess hemophilia A patient characteristics and reasons for switching from both patient/caregiver and physician perspectives. For this purpose, this research study will include hemophilia A patients who have switched from an existing therapy to Kovaltry or Jivi. In doing so, real world evidence will be obtained from both patient and physician perspectives offering key insights for effective therapeutic management of patients with hemophilia A and to more fully understand what drives patient switching from a patient perspective and a physician perspective.

DETAILED DESCRIPTION:
This observational study consists of a patient and a physician survey. This survey will consist of questions developed by Bayer and submitted to the Steering Committee of the existing registry, ATHN-2. Once enrolled to participate in the ATHN-2 registry and provided consent to participate in the Bayer nested study, patients who have switched from another product to Kovaltry or Jivi within the past 50 weeks or at the time of enrollment will be prompted to answer the additional survey questions.

Conclusion of the ATHN-2 registry is scheduled for 2021. Once data is cleaned and locked by the registry, the data will be delivered to Bayer for conduct of our analyses.

ELIGIBILITY:
Hemophilia A patients who have switched treatment to treatment with Kovaltry or Jivi within the past 50 weeks, who are enrolled the ATHN 2: Factor Switching Study, and who have consented to participate in the Kovaltry or Jivi specific module will be included in this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously treated hemophilia A patients enrolled into existing registry who have switched FVIII replacement treatment to Kovaltry or Jivi and provided consent to participate in the Bayer nested study
  ATHN's study with categorize selected subjects into two arms:
  * Arm A (Prospective): Patients who are switching factor replacement products and will be followed prospectively for 1 year post-switch
  * Arm B (Retrospective): Patients who have switched factor replacement products previously (within the past fifty weeks at the time of enrollments and will be followed prospectively until they reach a total of 52 weeks of observation. Historical data will be collected retrospectively for patients who switched prior to study entry.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Patient reported reasons for switching FVIII replacement treatment to Kovaltry or Jivi using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Patient expectations of switching FVIII replacement therapy to Kovaltry or Jivi would affect lifestyle/quality of life using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Patient expectations when adjusting to the new product after switch using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Patient reported root of expectations using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Patient reported reasons that would deter them from switching FVIII replacement products using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Physicians reported discipline using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Physicians reported reasons for switching FVIII replacement treatment to Kovaltry or Jivi using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Dosing Regimen (pre/post-switch) | Up to 4 years
  Data from consenting patients will be collected by ATHN
Physicians reported reason of newly selected dose/dosing interval using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Physicians reported rationale base for new dosing regimen selection using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Physicians reported communication about adjustment period when switching using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN
Physicians reported reasons that a provider would not encourage a patient to switch FVIII products using a Bayer designed survey | Up to 4 years
  Data from consenting patients will be collected by ATHN

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of California, San Diego, La Jolla, California
  - University of Colorado Denver Hemophilia and Thrombosis Center, Aurora, Colorado
  - Yale Hemophilia Treatment Center, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - St. Josephs Hemophilia Treatment Center, Tampa, Florida
  - Emory / Children's Healthcare of Atlanta, Atlanta, Georgia
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center IHTC, Indianapolis, Indiana
  - Louisiana Center for Bleeding and Clotting Disorders / Tulane, New Orleans, Louisiana
  - Maine Hemophilia and Thrombosis Center, Scarborough, Maine
  - The Johns Hopkins University Hemophilia Treatment Center, Baltimore, Maryland
  - Boston Hemophilia Center at Children's Hospital of Boston/Brigham Women's, Boston, Massachusetts
  - Univ of Michigan Hemophilia and Coagulation Disorders, Ann Arbor, Michigan
  - Michigan State University Center for Bleeding Disorders & Clotting Disorders, East Lansing, Michigan
  - Children's Mercy Hospital (Kansas City), Kansas City, Missouri
  - Dartmouth-Hitchcock Comprehensive Hemophilia and Thrombosis Center, Lebanon, New Hampshire
  - Weill Cornell Medicine, New York, New York
  - Mary M. Gooley Hemophilia Center, Inc., Rochester, New York
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Penn Comprehensive Hemophilia and Thrombophilia Program / Hospital UPENN, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern/Children's Health Dallas, Dallas, Texas
  - BloodWorks (Puget Sound), Seattle, Washington
  - Blood Center of Wisconsin, Inc. /Childrens Hosp of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field — http://clinicaltrials.bayer.com/